CLINICAL TRIAL: NCT06502210
Title: Identification of New Gene Spliceosomes in Neuroblastoma and Their Translational Application in Clinical Accurate Diagnosis and Therapy
Brief Title: Identification of New Gene Spliceosomes in Neuroblastoma
Status: Recruiting | Type: Observational
Sponsor: Affiliated Hospital of Nantong University (Other)
Responsible Party: Sponsor
Other Study IDs: LCYJ20242005
Record Dates: First submitted 2024-06-30; First posted 2024-07-16 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-04

CONDITIONS: Neuroblastoma
Keywords: Neuroblastoma; gene
MeSH Terms: conditions — Neuroblastoma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Biospecimen Retention: Samples With DNA — Researchers take neuroblastoma tissue and normal tissue adjacent to the tumor.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- neuroblastoma group: The resected tumor tissue of patients with neuroblastoma was taken by surgical operation as experimental group.
  Interventions: Procedure: Personalized surgical therapy of neuroblastoma
- Normal tissue adjacent to the tumor group: The normal tissue adjacent to tumor of patients with neuroblastoma was taken by surgical operation as control group.

INTERVENTIONS:
Procedure: Personalized surgical therapy of neuroblastoma — If the size of the tumor tissue is too large, the doctor gives the patient chemotherapy and then performs surgery to remove the tumor. In this study, the genotypes of children with neuroblastoma are screened by using Deep Sequencing Technology and Third Generation Sequencing Technology, and the treatment will be performed according to different therapeutic modalities.
  Groups: neuroblastoma group

SUMMARY:
Neuroblastoma is an early childhood embryonic malignancy that originates from neural crest cells. Neuroblastoma shows high heterogeneity in biological, morphological, genetic, and clinical features. At present, the main treatment methods for neuroblastoma are surgical treatment combined with chemotherapy after the operation and immunological therapy. However， clinical studies have found that 40%～50% of patients don't have good outcomes after postoperative chemotherapy.

The clinical trial study aims to screen the genotype of children with neuroblastoma and conduct an in-depth analysis of sequencing data and tumor-specific transcripts by using technologies--Deep Sequencing Technology and Third Generation Sequencing Technology.

The main questions this study aims to answer are： [Question 1]This study will use Third Generation Sequencing technology to find specific transcript variants associated with cancer differentiation; [Question 2]This study will identify possible tissue differential expression by using the Deep Sequencing Technology.

Participants will undergo surgery, during which doctors will remove tumor tissue and adjacent normal tissue. In this experiment, the tumor tissue of children with neuroblastoma will be used as the experimental group, and the adjacent normal tissue will be used as the control group. In this study， the different genotypes of children with neuroblastoma are screened by Deep Sequencing Technology and Third Generation Sequencing Technology. And according to the difference in genotypes， doctors will treat children with neuroblastoma personally. This study hopes to find new single nucleotide polymorphism and therapeutic targets.

DETAILED DESCRIPTION:
The clinical trial study aims to screen the genotype of children with neuroblastoma and conduct an in-depth analysis of sequencing data and tumor-specific transcripts using technologies--Deep Sequencing Technology and Third Generation Sequencing Technology. This study hopes to find new single nucleotide polymorphism and therapeutic targets.

Firstly, researchers collect tumor tissues and adjacent normal tissues of 20 children with neuroblastoma meeting the inclusion criteria and collect their clinical data. In this experiment, the tumor tissue of children with neuroblastoma will be used as the experimental group, and the adjacent normal tissue will be used as the control group.

Secondly, researchers will find differentially expressed genes using Deep Sequencing technology and Third Generation Sequencing Technology to sequence 7 neuroblastoma cell lines. The expression of the transcription isoforms was divided into one group of N-myc gene amplification and another group of N-myc gene non-amplification by using Third Generation Sequencing Technology. After extracting the total RNA from tissues, researchers check the RNA's purity, concentration, and integrity. If the RNA is tested up to standard, researchers will build a gene library. After the construction of the gene library is completed, researchers will use the machine to sequence tissues.

Finally, survival analysis and repeated measurements will be used to analyze the data of the experimental group and control group in this experiment. T-test will be used for measurement data. χ2 test will be used for counting data. Kaplan-Meier method and Cox regression analysis will be used for survival analysis. All statistical analyses will be performed using Statistical Analysis Software (Stata 26.0). P < 0.05 is considered significant.

ELIGIBILITY:
Inclusion Criteria:

* Children with neuroblastoma range in age from 0 to 14, regardless of gender;
* Preoperative imaging examinations indicate patient with neuroblastoma;
* Before postoperative chemotherapy, the patient's physical strength is good. At the same time, the results of white blood cells, neutrophils, hemoglobin, platelets, and other test indicators are all within normal range, which is in line with the treatment conditions of the relevant chemotherapy and immunotherapy;
* Preoperative pathological examination of the patient reveals neuroblastoma;
* Patients have no other history of malignant tumors;
* Patients voluntarily participate and sign informed consent and can comply with the study visit plan and other protocol requirements.

Exclusion Criteria:

* Patients who are found to have distant metastasis or ascites on preoperative examination are excluded;
* Patients with severe liver and kidney dysfunction, as well as those with autoimmune diseases are excluded;
* Patients with severe cardiovascular disease who can not tolerate general anesthesia are excluded;
* Patients who have other malignancies or blood disorders are excluded.

Ages: 1 Day to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The sample is from patients with neuroblastoma who underwent laparoscopic/open neuroblastoma surgery at Nantong University Affiliated Hospital from 2024 to 2026. Children with neuroblastoma range in age from 0 to 14, regardless of gender. Preoperative imaging examinations indicate a patient with neuroblastoma. Before postoperative chemotherapy, the patient's physical strength is good. A preoperative pathological examination of the patient reveals neuroblastoma. Patients have no other history of malignant tumors. Patients voluntarily participate and sign informed consent and can comply with the study visit plan and other protocol requirements.
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-08-31 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
The differential expression of tissue | 1 year
  The outcome measure is the change in tissue differential expression obtained by comparing the deep sequencing results of neuroblastoma tissue samples and normal tissue samples.
Specific transcript variant | 1 year
  The changes in tumor differentiation-related specific transcripts were found by comparing third-generation sequencing of neuroblastoma tissue sample cell lines.

CONTACTS AND LOCATIONS:
Overall Officials: Wenliang Ge, archiater, Study Chair — Nantong University Affiliated Hospital
Locations (1):
- Affiliated Hospital of Nantong University, Nantong, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pugh TJ, Morozova O, Attiyeh EF, Asgharzadeh S, Wei JS, Auclair D, Carter SL, Cibulskis K, Hanna M, Kiezun A, Kim J, Lawrence MS, Lichenstein L, McKenna A, Pedamallu CS, Ramos AH, Shefler E, Sivachenko A, Sougnez C, Stewart C, Ally A, Birol I, Chiu R, Corbett RD, Hirst M, Jackman SD, Kamoh B, Khodabakshi AH, Krzywinski M, Lo A, Moore RA, Mungall KL, Qian J, Tam A, Thiessen N, Zhao Y, Cole KA, Diamond M, Diskin SJ, Mosse YP, Wood AC, Ji L, Sposto R, Badgett T, London WB, Moyer Y, Gastier-Foster JM, Smith MA, Guidry Auvil JM, Gerhard DS, Hogarty MD, Jones SJ, Lander ES, Gabriel SB, Getz G, Seeger RC, Khan J, Marra MA, Meyerson M, Maris JM. The genetic landscape of high-risk neuroblastoma. Nat Genet. 2013 Mar;45(3):279-84. doi: 10.1038/ng.2529. Epub 2013 Jan 20. PMID 23334666
- [Background] Schramm A, Koster J, Assenov Y, Althoff K, Peifer M, Mahlow E, Odersky A, Beisser D, Ernst C, Henssen AG, Stephan H, Schroder C, Heukamp L, Engesser A, Kahlert Y, Theissen J, Hero B, Roels F, Altmuller J, Nurnberg P, Astrahantseff K, Gloeckner C, De Preter K, Plass C, Lee S, Lode HN, Henrich KO, Gartlgruber M, Speleman F, Schmezer P, Westermann F, Rahmann S, Fischer M, Eggert A, Schulte JH. Mutational dynamics between primary and relapse neuroblastomas. Nat Genet. 2015 Aug;47(8):872-7. doi: 10.1038/ng.3349. Epub 2015 Jun 29. PMID 26121086
- [Background] Lopez G, Conkrite KL, Doepner M, Rathi KS, Modi A, Vaksman Z, Farra LM, Hyson E, Noureddine M, Wei JS, Smith MA, Asgharzadeh S, Seeger RC, Khan J, Guidry Auvil J, Gerhard DS, Maris JM, Diskin SJ. Somatic structural variation targets neurodevelopmental genes and identifies SHANK2 as a tumor suppressor in neuroblastoma. Genome Res. 2020 Sep;30(9):1228-1242. doi: 10.1101/gr.252106.119. Epub 2020 Aug 13. PMID 32796005
- [Background] Brady SW, Liu Y, Ma X, Gout AM, Hagiwara K, Zhou X, Wang J, Macias M, Chen X, Easton J, Mulder HL, Rusch M, Wang L, Nakitandwe J, Lei S, Davis EM, Naranjo A, Cheng C, Maris JM, Downing JR, Cheung NV, Hogarty MD, Dyer MA, Zhang J. Pan-neuroblastoma analysis reveals age- and signature-associated driver alterations. Nat Commun. 2020 Oct 14;11(1):5183. doi: 10.1038/s41467-020-18987-4. PMID 33056981
- [Background] Qiu B, Matthay KK. Advancing therapy for neuroblastoma. Nat Rev Clin Oncol. 2022 Aug;19(8):515-533. doi: 10.1038/s41571-022-00643-z. Epub 2022 May 25. PMID 35614230
- [Background] Rickman DS, Schulte JH, Eilers M. The Expanding World of N-MYC-Driven Tumors. Cancer Discov. 2018 Feb;8(2):150-163. doi: 10.1158/2159-8290.CD-17-0273. Epub 2018 Jan 22. PMID 29358508
- [Background] Otte J, Dyberg C, Pepich A, Johnsen JI. MYCN Function in Neuroblastoma Development. Front Oncol. 2021 Jan 27;10:624079. doi: 10.3389/fonc.2020.624079. eCollection 2020. PMID 33585251
- [Background] Zimmerman MW, Liu Y, He S, Durbin AD, Abraham BJ, Easton J, Shao Y, Xu B, Zhu S, Zhang X, Li Z, Weichert-Leahey N, Young RA, Zhang J, Look AT. MYC Drives a Subset of High-Risk Pediatric Neuroblastomas and Is Activated through Mechanisms Including Enhancer Hijacking and Focal Enhancer Amplification. Cancer Discov. 2018 Mar;8(3):320-335. doi: 10.1158/2159-8290.CD-17-0993. Epub 2017 Dec 28. PMID 29284669
- [Background] Rosswog C, Fassunke J, Ernst A, Schomig-Markiefka B, Merkelbach-Bruse S, Bartenhagen C, Cartolano M, Ackermann S, Theissen J, Blattner-Johnson M, Jones B, Schramm K, Altmuller J, Nurnberg P, Ortmann M, Berthold F, Peifer M, Buttner R, Westermann F, Schulte JH, Simon T, Hero B, Fischer M. Genomic ALK alterations in primary and relapsed neuroblastoma. Br J Cancer. 2023 Apr;128(8):1559-1571. doi: 10.1038/s41416-023-02208-y. Epub 2023 Feb 17. PMID 36807339
- [Background] Bellini A, Potschger U, Bernard V, Lapouble E, Baulande S, Ambros PF, Auger N, Beiske K, Bernkopf M, Betts DR, Bhalshankar J, Bown N, de Preter K, Clement N, Combaret V, Font de Mora J, George SL, Jimenez I, Jeison M, Marques B, Martinsson T, Mazzocco K, Morini M, Muhlethaler-Mottet A, Noguera R, Pierron G, Rossing M, Taschner-Mandl S, Van Roy N, Vicha A, Chesler L, Balwierz W, Castel V, Elliott M, Kogner P, Laureys G, Luksch R, Malis J, Popovic-Beck M, Ash S, Delattre O, Valteau-Couanet D, Tweddle DA, Ladenstein R, Schleiermacher G. Frequency and Prognostic Impact of ALK Amplifications and Mutations in the European Neuroblastoma Study Group (SIOPEN) High-Risk Neuroblastoma Trial (HR-NBL1). J Clin Oncol. 2021 Oct 20;39(30):3377-3390. doi: 10.1200/JCO.21.00086. Epub 2021 Jun 11. PMID 34115544
- [Background] Schulte JH, Eggert A. ALK Inhibitors in Neuroblastoma: A Sprint from Bench to Bedside. Clin Cancer Res. 2021 Jul 1;27(13):3507-3509. doi: 10.1158/1078-0432.CCR-21-0627. Epub 2021 May 4. PMID 33947691
- [Background] D'Oto A, Fang J, Jin H, Xu B, Singh S, Mullasseril A, Jones V, Abu-Zaid A, von Buttlar X, Cooke B, Hu D, Shohet J, Murphy AJ, Davidoff AM, Yang J. KDM6B promotes activation of the oncogenic CDK4/6-pRB-E2F pathway by maintaining enhancer activity in MYCN-amplified neuroblastoma. Nat Commun. 2021 Dec 10;12(1):7204. doi: 10.1038/s41467-021-27502-2. PMID 34893606
- [Background] Aygun N. Biological and Genetic Features of Neuroblastoma and Their Clinical Importance. Curr Pediatr Rev. 2018;14(2):73-90. doi: 10.2174/1573396314666180129101627. PMID 29380702
- [Background] Yue ZX, Xing TY, Zhao W, Zhao Q, Wang XS, Su Y, Gao C, Liu SG, Ma XL. MYCN amplification plus 1p36 loss of heterozygosity predicts ultra high risk in bone marrow metastatic neuroblastoma. Cancer Med. 2022 Apr;11(8):1837-1849. doi: 10.1002/cam4.4583. Epub 2022 Feb 9. PMID 35137546
- [Background] Garcia-Lopez J, Wallace K, Otero JH, Olsen R, Wang YD, Finkelstein D, Gudenas BL, Rehg JE, Northcott P, Davidoff AM, Freeman KW. Large 1p36 Deletions Affecting Arid1a Locus Facilitate Mycn-Driven Oncogenesis in Neuroblastoma. Cell Rep. 2020 Jan 14;30(2):454-464.e5. doi: 10.1016/j.celrep.2019.12.048. PMID 31940489
- [Background] Valentijn LJ, Koster J, Zwijnenburg DA, Hasselt NE, van Sluis P, Volckmann R, van Noesel MM, George RE, Tytgat GA, Molenaar JJ, Versteeg R. TERT rearrangements are frequent in neuroblastoma and identify aggressive tumors. Nat Genet. 2015 Dec;47(12):1411-4. doi: 10.1038/ng.3438. Epub 2015 Nov 2. PMID 26523776
- [Background] Molenaar JJ, Koster J, Zwijnenburg DA, van Sluis P, Valentijn LJ, van der Ploeg I, Hamdi M, van Nes J, Westerman BA, van Arkel J, Ebus ME, Haneveld F, Lakeman A, Schild L, Molenaar P, Stroeken P, van Noesel MM, Ora I, Santo EE, Caron HN, Westerhout EM, Versteeg R. Sequencing of neuroblastoma identifies chromothripsis and defects in neuritogenesis genes. Nature. 2012 Feb 22;483(7391):589-93. doi: 10.1038/nature10910. PMID 22367537
- [Background] Verhaak RGW, Bafna V, Mischel PS. Extrachromosomal oncogene amplification in tumour pathogenesis and evolution. Nat Rev Cancer. 2019 May;19(5):283-288. doi: 10.1038/s41568-019-0128-6. PMID 30872802
- [Background] Koche RP, Rodriguez-Fos E, Helmsauer K, Burkert M, MacArthur IC, Maag J, Chamorro R, Munoz-Perez N, Puiggros M, Dorado Garcia H, Bei Y, Roefzaad C, Bardinet V, Szymansky A, Winkler A, Thole T, Timme N, Kasack K, Fuchs S, Klironomos F, Thiessen N, Blanc E, Schmelz K, Kunkele A, Hundsdorfer P, Rosswog C, Theissen J, Beule D, Deubzer H, Sauer S, Toedling J, Fischer M, Hertwig F, Schwarz RF, Eggert A, Torrents D, Schulte JH, Henssen AG. Extrachromosomal circular DNA drives oncogenic genome remodeling in neuroblastoma. Nat Genet. 2020 Jan;52(1):29-34. doi: 10.1038/s41588-019-0547-z. Epub 2019 Dec 16. PMID 31844324
- [Background] Helmsauer K, Valieva ME, Ali S, Chamorro Gonzalez R, Schopflin R, Roefzaad C, Bei Y, Dorado Garcia H, Rodriguez-Fos E, Puiggros M, Kasack K, Haase K, Keskeny C, Chen CY, Kuschel LP, Euskirchen P, Heinrich V, Robson MI, Rosswog C, Toedling J, Szymansky A, Hertwig F, Fischer M, Torrents D, Eggert A, Schulte JH, Mundlos S, Henssen AG, Koche RP. Enhancer hijacking determines extrachromosomal circular MYCN amplicon architecture in neuroblastoma. Nat Commun. 2020 Nov 16;11(1):5823. doi: 10.1038/s41467-020-19452-y. PMID 33199677
- [Background] Paolini L, Hussain S, Galardy PJ. Chromosome instability in neuroblastoma: A pathway to aggressive disease. Front Oncol. 2022 Oct 20;12:988972. doi: 10.3389/fonc.2022.988972. eCollection 2022. PMID 36338721
- [Background] De Bernardi B, Di Cataldo A, Garaventa A, Massirio P, Viscardi E, Podda MG, Castellano A, D'Angelo P, Tirtei E, Melchionda F, Vetrella S, De Leonardis F, D'Ippolito C, Tondo A, Nonnis A, Erminio G, Gigliotti AR, Mazzocco K, Haupt R. Stage 4 s neuroblastoma: features, management and outcome of 268 cases from the Italian Neuroblastoma Registry. Ital J Pediatr. 2019 Jan 11;45(1):8. doi: 10.1186/s13052-018-0599-1. PMID 30634996
- [Background] Janoueix-Lerosey I, Schleiermacher G, Michels E, Mosseri V, Ribeiro A, Lequin D, Vermeulen J, Couturier J, Peuchmaur M, Valent A, Plantaz D, Rubie H, Valteau-Couanet D, Thomas C, Combaret V, Rousseau R, Eggert A, Michon J, Speleman F, Delattre O. Overall genomic pattern is a predictor of outcome in neuroblastoma. J Clin Oncol. 2009 Mar 1;27(7):1026-33. doi: 10.1200/JCO.2008.16.0630. Epub 2009 Jan 26. PMID 19171713
- [Background] Schleiermacher G, Janoueix-Lerosey I, Ribeiro A, Klijanienko J, Couturier J, Pierron G, Mosseri V, Valent A, Auger N, Plantaz D, Rubie H, Valteau-Couanet D, Bourdeaut F, Combaret V, Bergeron C, Michon J, Delattre O. Accumulation of segmental alterations determines progression in neuroblastoma. J Clin Oncol. 2010 Jul 1;28(19):3122-30. doi: 10.1200/JCO.2009.26.7955. Epub 2010 Jun 1. PMID 20516441
- [Background] Ackermann S, Cartolano M, Hero B, Welte A, Kahlert Y, Roderwieser A, Bartenhagen C, Walter E, Gecht J, Kerschke L, Volland R, Menon R, Heuckmann JM, Gartlgruber M, Hartlieb S, Henrich KO, Okonechnikov K, Altmuller J, Nurnberg P, Lefever S, de Wilde B, Sand F, Ikram F, Rosswog C, Fischer J, Theissen J, Hertwig F, Singhi AD, Simon T, Vogel W, Perner S, Krug B, Schmidt M, Rahmann S, Achter V, Lang U, Vokuhl C, Ortmann M, Buttner R, Eggert A, Speleman F, O'Sullivan RJ, Thomas RK, Berthold F, Vandesompele J, Schramm A, Westermann F, Schulte JH, Peifer M, Fischer M. A mechanistic classification of clinical phenotypes in neuroblastoma. Science. 2018 Dec 7;362(6419):1165-1170. doi: 10.1126/science.aat6768. PMID 30523111
- [Background] Peifer M, Hertwig F, Roels F, Dreidax D, Gartlgruber M, Menon R, Kramer A, Roncaioli JL, Sand F, Heuckmann JM, Ikram F, Schmidt R, Ackermann S, Engesser A, Kahlert Y, Vogel W, Altmuller J, Nurnberg P, Thierry-Mieg J, Thierry-Mieg D, Mariappan A, Heynck S, Mariotti E, Henrich KO, Gloeckner C, Bosco G, Leuschner I, Schweiger MR, Savelyeva L, Watkins SC, Shao C, Bell E, Hofer T, Achter V, Lang U, Theissen J, Volland R, Saadati M, Eggert A, de Wilde B, Berthold F, Peng Z, Zhao C, Shi L, Ortmann M, Buttner R, Perner S, Hero B, Schramm A, Schulte JH, Herrmann C, O'Sullivan RJ, Westermann F, Thomas RK, Fischer M. Telomerase activation by genomic rearrangements in high-risk neuroblastoma. Nature. 2015 Oct 29;526(7575):700-4. doi: 10.1038/nature14980. Epub 2015 Oct 14. PMID 26466568
- [Background] Roderwieser A, Sand F, Walter E, Fischer J, Gecht J, Bartenhagen C, Ackermann S, Otte F, Welte A, Kahlert Y, Lieberz D, Hertwig F, Reinhardt HC, Simon T, Peifer M, Ortmann M, Buttner R, Hero B, O'Sullivan RJ, Berthold F, Fischer M. Telomerase Is a Prognostic Marker of Poor Outcome and a Therapeutic Target in Neuroblastoma. JCO Precis Oncol. 2019 Dec;3:1-20. doi: 10.1200/PO.19.00072. PMID 35100718
- [Background] Yu EY, Zahid SS, Aloe S, Falck-Pedersen E, Zhou XK, Cheung NV, Lue NF. Reciprocal impacts of telomerase activity and ADRN/MES differentiation state in neuroblastoma tumor biology. Commun Biol. 2021 Nov 19;4(1):1315. doi: 10.1038/s42003-021-02821-8. PMID 34799676
- [Background] Hartlieb SA, Sieverling L, Nadler-Holly M, Ziehm M, Toprak UH, Herrmann C, Ishaque N, Okonechnikov K, Gartlgruber M, Park YG, Wecht EM, Savelyeva L, Henrich KO, Rosswog C, Fischer M, Hero B, Jones DTW, Pfaff E, Witt O, Pfister SM, Volckmann R, Koster J, Kiesel K, Rippe K, Taschner-Mandl S, Ambros P, Brors B, Selbach M, Feuerbach L, Westermann F. Alternative lengthening of telomeres in childhood neuroblastoma from genome to proteome. Nat Commun. 2021 Feb 24;12(1):1269. doi: 10.1038/s41467-021-21247-8. PMID 33627664
- [Background] Cheung NK, Zhang J, Lu C, Parker M, Bahrami A, Tickoo SK, Heguy A, Pappo AS, Federico S, Dalton J, Cheung IY, Ding L, Fulton R, Wang J, Chen X, Becksfort J, Wu J, Billups CA, Ellison D, Mardis ER, Wilson RK, Downing JR, Dyer MA; St Jude Children's Research Hospital-Washington University Pediatric Cancer Genome Project. Association of age at diagnosis and genetic mutations in patients with neuroblastoma. JAMA. 2012 Mar 14;307(10):1062-71. doi: 10.1001/jama.2012.228. PMID 22416102
- [Background] Qadeer ZA, Valle-Garcia D, Hasson D, Sun Z, Cook A, Nguyen C, Soriano A, Ma A, Griffiths LM, Zeineldin M, Filipescu D, Jubierre L, Chowdhury A, Deevy O, Chen X, Finkelstein DB, Bahrami A, Stewart E, Federico S, Gallego S, Dekio F, Fowkes M, Meni D, Maris JM, Weiss WA, Roberts SS, Cheung NV, Jin J, Segura MF, Dyer MA, Bernstein E. ATRX In-Frame Fusion Neuroblastoma Is Sensitive to EZH2 Inhibition via Modulation of Neuronal Gene Signatures. Cancer Cell. 2019 Nov 11;36(5):512-527.e9. doi: 10.1016/j.ccell.2019.09.002. Epub 2019 Oct 17. PMID 31631027
- [Background] George SL, Parmar V, Lorenzi F, Marshall LV, Jamin Y, Poon E, Angelini P, Chesler L. Novel therapeutic strategies targeting telomere maintenance mechanisms in high-risk neuroblastoma. J Exp Clin Cancer Res. 2020 May 6;39(1):78. doi: 10.1186/s13046-020-01582-2. PMID 32375866

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-01-05): https://cdn.clinicaltrials.gov/large-docs/10/NCT06502210/Prot_SAP_000.pdf